CLINICAL TRIAL: NCT06760377
Title: Dietary Supplements for Reduction of Intestinal Permeability Levels
Acronym: permeability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Isidro Fernández López, Principal investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UComplutenseMadrid Intestinal
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Intestinal Permeability; Leaky Gut Syndrome; Zonulin
Keywords: intestinal permeability; leaky gut syndrome; zonulin; tight junctions

STUDY DESIGN:
Intervention Model Description: It has been estimated to conduct a trial with subjects who are distributed in two groups: an intervention group of patients to whom supplementation is provided, and a control group of subjects who do not receive any type of supplementation.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement Group (Experimental): Subjects belonging to the experimental group will be provided with the PermeaIntest supplement, which they will take for 60 days, 1 sachet in the morning and 1 sachet in the evening in half a glass of water. Subjects will have a stool sample collected before and after ingestion of the dietary supplement.
  Interventions: Dietary Supplement: Dietary supplement Group
- Control group (No Intervention): A control group of subjects not receiving any type of supplementation will be used to compare the effectiveness of the treatment. Subjects will have a stool sample collected before and after a period of 60 days

INTERVENTIONS:
Dietary Supplement: Dietary supplement Group — Subjects belonging to the experimental group will be provided with the PermeaIntest supplement, which they will take for 60 days, 1 sachet in the morning and 1 sachet in the evening in half a glass of water. Subjects will have a stool sample collected before and after ingestion of the dietary supplement.
  Arms: Dietary supplement Group

SUMMARY:
A randomised and controlled trial, in which the effect of a dietary supplement is evaluated for reduction of intestinal permeability levels of subjects with high levels of zonulin in feces

DETAILED DESCRIPTION:
Randomized clinical trial, with masking of the statistician and the evaluator, to assess the effect of a food supplement, composed of substances that promote intestinal mucosa repair, on the levels of zonulin in feces and consequently on intestinal permeability. A control group of subjects not receiving any type of supplementation will be used to compare the effectiveness of the treatment.

The main objective of this study is to determine if the use of a dietary supplement composed of glutamine, butyrate and lion's mane, among others, corrects the levels of zonulin in feces.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 65 years of age with elevated levels of zonulin in stool (greater than 80 ng/ml).

Exclusion Criteria:

* Taking any type of antibiotic in the last month
* Taking prebiotics or probiotics products in the last month.
* Taking laxatives in the last month.
* Undergoing any medicinal treatment
* Pregnancy
* Subject with a history of current gastrointestinal pathology or disorder such as: acute colon pathology, acute haemorrhagic colitis, suspected digestive perforation, recent abdominal surgery, severe arterial hypertension, abdominal hernia, colon neoplasia, history of cardiac syncope, renal failure, liver cirrhosis, epilepsy, severe psychiatric illness (psychosis), necrosis due to abdominal irradiation, severe anaemia, severe neurovegetative lability.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Zonulin levels in feces | 60 days
  Zonulin levels in feces, assessed in ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fasano A, Shea-Donohue T. Mechanisms of disease: the role of intestinal barrier function in the pathogenesis of gastrointestinal autoimmune diseases. Nat Clin Pract Gastroenterol Hepatol. 2005 Sep;2(9):416-22. doi: 10.1038/ncpgasthep0259. PMID 16265432
- [Result] Fasano A. Regulation of intercellular tight junctions by zonula occludens toxin and its eukaryotic analogue zonulin. Ann N Y Acad Sci. 2000;915:214-22. doi: 10.1111/j.1749-6632.2000.tb05244.x. PMID 11193578
- [Result] Lerner A, Matthias T. Changes in intestinal tight junction permeability associated with industrial food additives explain the rising incidence of autoimmune disease. Autoimmun Rev. 2015 Jun;14(6):479-89. doi: 10.1016/j.autrev.2015.01.009. Epub 2015 Feb 9. PMID 25676324
- [Result] Fasano A. Zonulin and its regulation of intestinal barrier function: the biological door to inflammation, autoimmunity, and cancer. Physiol Rev. 2011 Jan;91(1):151-75. doi: 10.1152/physrev.00003.2008. PMID 21248165
- [Result] Tripathi A, Lammers KM, Goldblum S, Shea-Donohue T, Netzel-Arnett S, Buzza MS, Antalis TM, Vogel SN, Zhao A, Yang S, Arrietta MC, Meddings JB, Fasano A. Identification of human zonulin, a physiological modulator of tight junctions, as prehaptoglobin-2. Proc Natl Acad Sci U S A. 2009 Sep 29;106(39):16799-804. doi: 10.1073/pnas.0906773106. Epub 2009 Sep 15. PMID 19805376